CLINICAL TRIAL: NCT06426303
Title: Sex Differences in Trauma, Inflammation and Brain Function and the Implications for Treatment Efficacy in Alcohol Use Disorder
Acronym: ABSTAIN
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Milky Kohno (Other)
Collaborators: Portland VA Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, Milky Kohno, Assistant Professor, Oregon Health and Science University
Organization: Oregon Health and Science University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 25536
Record Dates: First submitted 2024-04-19; First posted 2024-05-23 (Actual); Last update posted 2024-07-18 (Actual); Status verified 2024-07

CONDITIONS: Alcohol Use Disorder
Keywords: Naltrexone
MeSH Terms: conditions — Alcoholism | interventions — Naltrexone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Alcohol Use Disorder (AUD) (Experimental): Drug: Naltrexone Half of the study participants with AUD will take an oral tablet of 50 mg naltrexone once daily for one week followed by 11 weeks of 100 mg naltrexone orally, once daily.
  Drug: Placebo oral tablet The other half of study participants will receive an identical looking placebo in tablet form and take the medication using an identical schedule as the real drug.
  Drug type will be randomized.
  Interventions: Drug: Naltrexone
- Healthy Controls (No Intervention): Baseline measures will be taken but controls will not continue to the drug trial.

INTERVENTIONS:
Drug: Naltrexone — 12-week randomized double blinded placebo-controlled drug trial titrating drug/placebo dose after 1 week.
  Other Names: Revia
  Arms: Alcohol Use Disorder (AUD)

SUMMARY:
The goal of this clinical trial is to identify sex-specific biomarkers that confer greater susceptibility for Alcohol Use Disorder (AUD) and differentiate how treatment response varies by sex in people with Alcohol Use Disorder.

The main questions it aims to answer are:

* How does trauma affect emotion regulation, inflammation, and limbic function, and what are the sex-dependent effects of NTX (Naltrexone) on these aspects?
* What is the mechanism of Naltrexone (NTX), and how does it potentially moderate reductions in alcohol use through changes in or interactions between emotion regulation, inflammation, or limbic system function?

Participants will

* Be consented and will undergo comprehensive screening for eligibility criteria
* Complete behavioral assessments and neuropsychological assessments, as well as neurocognitive assessments and neuroimaging measures
* Provide urine samples for a urine drug screen (UDS) and urine pregnancy test (for women), and have blood and a cheek swab collected and stored in the repository
* Take a study drug once daily for 12 weeks and track drug usage and effects in a study journal
* Undergo weekly assessment calls and bi-weekly medical follow-up safety exams

Researchers will compare naltrexone to placebo in AUD to see if naltrexone is effective in reducing alcohol cravings and promoting abstinence.

Researchers will also compare baseline measures between AUD and Healthy Controls.

DETAILED DESCRIPTION:
A twelve-week randomized placebo-controlled trial of naltrexone (NTX) will be conducted in one hundred people with alcohol use disorder (AUD), fifty of which will be women. Fifty healthy participants will serve as controls for baseline measures. We will use validated measures to comprehensively assess trauma exposure including: military sexual trauma (MST), physical or sexual assault, combat exposure, intimate partner violence, and other traumatic events. Emotion regulation will be assessed with the Cognitive Emotion Regulation questionnaire and Difficulty in Emotion Regulation scale. Functional magnetic resonance imaging at rest and during an emotion regulation task will assess limbic system connectivity and reactivity. Inflammation will be indexed with a multiplex panel assay of peripheral inflammatory markers. Days of alcohol use and average weekly standard drinks will be assessed at each time-point.

ELIGIBILITY:
Inclusion Criteria:

* 18-60 years old
* Veteran enrolled in VHA healthcare

Alcohol Group:

* must meet diagnosis for recent alcohol-use disorder (DSM-V)
* willing to return for follow-up visits and can participate for 12-weeks

Control Group:

* must not meet DSM-V criteria for a use disorder other than nicotine

Exclusion Criteria:

* Clinically significant neurological, endocrine, hepatic, or systemic disease that would compromise safe participation or confound outcomes
* Left-handedness
* Axis-1 psychiatric diagnoses other than anxiety, depression or post-traumatic stress disorder
* Recreational or prescriptive use of psychotropic medications
* Recreational or prescriptive use of opioid medications or have a past or current history of abuse or dependence on opioids
* MRI contraindications (e.g. metal in body)
* Positive urine drug screen, except for nicotine and marijuana, on test days
* Women who are pregnant or breastfeeding
* Participants on hormonal therapy or treatments other than pregnancy contraceptives
* Autoimmune or neurodegenerative diseases that present with neuroinflammation (multiple sclerosis, amyotrophic lateral sclerosis, Alzheimer's, Parkinson's)
* Current participation in an investigational drug study
* Alcohol group: < 5 days and > 3 weeks of abstinence from alcohol
* Alcohol group: Liver disease requiring medication or medical treatment, and/or aspartate or alanine aminotransferase levels greater than 3 times the upper limit of normal, gastrointestinal or renal disease that would significantly impair absorption, metabolism or excretion of study drug, or require medical treatment.
* Non-english speaker

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-05-02 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in alcohol use (number of drinking days, amount used per day) | Baseline and Week 12
  Drinking days and average number of weekly standard drinks will be measured at baseline and at follow-up
Changes from baseline in peripheral immune biomarkers associated with inflammation | Baseline and Week 12
  Plasma samples will be analyzed using a customized, high-sensitivity magnetic bead multiplex assay Luminex system. Samples will be prepared and analyzed to measure peripheral immune markers: interleukin (IL)-1-beta, IL-6, IL-10, tumor necrosis factor (TNF)-alpha, brain-derived neurotrophic factor (BDNF), monocyte chemotactic protein (MCP)-1 and neural cell adhesion molecule (NCAM). Intra-and inter-assay coefficients of variation, as indices of within-and between-assay precision, respectively, will be calculated to examine the reliability of cytokine measurements.
Changes in limbic functional connectivity | Baseline and Week 12
  Resting-state functional magnetic resonance imaging (rs-fMRI) will be used to assess changes in limbic system connectivity. Correlation coefficients of low-frequency oscillations in the fMRI blood oxygenation level dependent (BOLD) signal between regions and between large-scale resting-state networks in the brain will be z-score transformed. A score of 0 indicates no change while higher or lower scores indicate increased or decreased connectivity, respectively.
Changes from baseline in BOLD signal brain activation during an emotion regulation fMRI task | Baseline and Week 12
  The task will assess emotional reactivity and regulation to negative and stressful images. Each event (cue, neutral-look, negative-look, negative-reappraise and rating scale of negative affect) will be modeled using a canonical hemodynamic response function with a time derivative. The contrasts of interest will be Negative-look vs Neutral-look and Negative-look vs Negative-reappraise. Amygdala BOLD signal estimates will be extracted to calculate percent-change.
Changes from baseline in emotion regulation assessed with the Difficulty in Emotion Regulation Scale (DERS) | Baseline and Week 12
  DERS is a 36-item self-report questionnaire scored on a 5-point scale from 1 (almost never) to 5 (almost always), with total score ranging from 36 to 180. It measures emotion regulation difficulties across six dimensions: 1. Non-acceptance of emotional responses, 2. Difficulties engaging in goal-directed behavior, 3. Impulse control difficulties, 4. Lack of emotional awareness, 5. Limited access to effective emotion regulation strategies, 6. Lack of emotional clarity. Higher scores suggest greater difficulties in emotion regulation.
Changes from baseline in emotion regulation assessed with the Cognitive Emotion Regulation Questionnaire (CERQ) | Baseline and Week 12
  CERQ is a 36-item self-report questionnaire that identifies cognitive emotion regulation or cognitive coping strategies used after having experienced negative events or situations. Scores can identify individual strategies to compare with normed scores from various populations. The nine cognitive emotion regulation strategies are measured on a 5-point Likert scale ranging from 1 to 5, with scores being obtained by calculating the mean scores belonging to a particular subscale. Higher subscale scores indicate greater use of a specific cognitive strategy.

SECONDARY OUTCOMES:
Change from baseline in craving (include craving measures/questionnaires) | Baseline and Week 12
  The Brief Alcohol Craving Scale, a 10-item self-report assessment of craving, will be used. Participants will be prompted with a statement regarding alcohol cravings and will choose an answer ranging between "strongly disagree" and "strongly agree."
Differences in baseline trauma exposure (composite score) | Baseline and Week 12
  Department of Veterans Affairs Military Sexual Trauma Screening consists of two questions used nationally within the Veterans Heath Administration (VHA) to screen for MST. Response options are yes, no, or decline to respond.
  Trauma Assessment for Adults (TAA) is a 17-item self-report on combat exposure, physical or sexual assault, surviving serious accidents and other threatening life events.
  Life Stressor Checklist-Revised (LSC-R) includes self-report measures relevant to women such as abortion or caregiver duties, in addition to 30 life events related to natural disasters, physical or sexual assault, death of a relative, incarceration and financial hardships.
  Childhood Maltreatment questionnaire is 70 items in five dimensions: emotional, physical, and sexual abuse, and physical and emotional neglect. A 7-point scale will be used to indicate level of trauma
Change from baseline in neuropsychological testing scores | Baseline and Week 12
  The Standard Neuropsychological Battery will be used

CONTACTS AND LOCATIONS:
Locations (1):
- VA Portland Health Care System, Portland, Oregon, United States